CLINICAL TRIAL: NCT05890560
Title: Comparison of the Two-year Efficacy of Three Exercise Rehabilitation Strategies on Dyspnea in Patients Who Presented With Secondary Respiratory Distress Syndrome Secondary to Severe COVID-19 Pneumonia
Brief Title: Two-year Efficacy of Three Exercise Rehabilitation Strategies on Dyspnea in Patients Who Presented With Secondary Respiratory Distress Syndrome Secondary to Severe COVID-19 Pneumonia
Acronym: RECOVER_FU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RECOVER_FollowUp
Record Dates: First submitted 2023-06-05; First posted 2023-06-06 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Dyspnea; COVID-19
MeSH Terms: conditions — Dyspnea; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dyspnea is defined by a subjective sensation of respiratory discomfort, the intensity of which varies according to the terrain, the anamnesis and the cause. Resuscitation is associated with many causes of dyspnea, including initial distress, mechanical ventilation, or after-effects following the pathology and its management.

Respiratory distress is the most severe form of impaired lung function. It is the first cause of hospitalization in intensive care. This distress, indicative of the failure of the respiratory system, is always severe and potentially fatal. It therefore constitutes an absolute therapeutic emergency. Dyspnea is often the revealing symptom of the condition and the urgency surrounding its management is an additional factor of concern for the patient. As a result, dyspnea is a pejorative element associated with severity or even death.

In patients surviving the initial condition, dyspnea persists and can be found months or even years later, despite the initial rehabilitation. It is strongly associated with anxiety or even the fear of dying and contributes to the occurrence of post-traumatic stress syndromes. This persistent sensation of respiratory discomfort, limiting the patient's autonomy in his activities of daily living, seems to be able to reduce his quality of life. In addition, the perpetuation of this dyspnea could favor a spiral of deconditioning causing a progressive deterioration of the cardio-respiratory system justifying new hospitalizations.

In patients with chronic respiratory failure, exercise rehabilitation supervised by hysiotherapists allows, in addition to improving autonomy, a significant reduction in dyspnoea, thus increasing the quality of life of these patients.

The main objective of this study is to evaluate the effect at 2 years of 3 modes of management of dyspnea: exercise rehabilitation, standard physiotherapy and "usual care" on post-resuscitation dyspnea in patients with presented with severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Patients in the RECOVER study (NCTT04569266):

* Patient ≥ 18 years old
* Patient meeting the inclusion criteria for this study (see appendix 1)
* Patient more than 2 years from their release from intensive care
* French-speaking patient
* Patient not objecting to their participation in this research

Usual care patients

* Patient ≥ 18 years old
* Patient having presented a respiratory infection by SARS-Cov-2 confirmed biologically in the laboratory by PCR or any other commercial or public health test or diagnosed by CT scan
* Patient who was under invasive mechanical ventilation during a stay in intensive care in the center of Versailles for more than 48 consecutive hours following infection by SARS-Cov-2 between 01/03/2020 and 26/01/2022
* Patient more than 2 years from their release from intensive care
* French-speaking patient
* Patient not objecting to their participation in this research

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who was under invasive mechanical ventilation during a stay in intensive care in the center of Versailles for more than 48 consecutive hours following infection by SARS-Cov-2 between 01/03/2020 and 26/01/2022, more than 2 years from their release from intensive care
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of exercise rehabilitation on post-ICU dyspnea | Year 2
  This outcome corresponds to the comparison of Multidimensional Dyspnea Profile (MDP) scale assessment of dyspnea between year 2 and Day 1. The Multidimensional Dyspnea Profile (MDP) assesses overall breathing discomfort, sensory qualities, and emotional responses in laboratory and clinical settings. The MDP consist of 11 descriptors of breathlessness rated using numerical rating scales (NRS) ranging from 0 to 10. A total score can be summarised as well as an immediate perception subdomain (6 items), and an emotional response subdomain (5 items).

SECONDARY OUTCOMES:
Evaluate the effect of exercise rehabilitation on functional dyspnea | Year2
  This outcome corresponds to the comparison of dyspnea on the Modified Medical Research Council (mMRC) scale between year 2 and day1. The mMRC (Modified Medical Research Council) Dyspnoea Scale is used to assess the degree of baseline functional disability due to dyspnoea. It is useful in characterising baseline dyspnoea in patients.
Evaluate the effect of stress rehabilitation on quality of life at the end of exercise rehabilitation | Year2
  This outcome corresponds to the comparison of Short-Form Quality of Life Assessment (SF-36) at the end of exercise rehabilitation (Year2 by comparison day 1).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe ROMANET, Study Director — Fondation Hôpital Saint-Joseph
Locations (4):
- France (4):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Fondation Hôpital Saint-Joseph, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier André Mignot, Versailles

REFERENCES:
- [Background] Romanet C, Wormser J, Fels A, Lucas P, Prudat C, Sacco E, Bruel C, Plantefeve G, Pene F, Chatellier G, Philippart F. Effectiveness of exercise training on the dyspnoea of individuals with long COVID: A randomised controlled multicentre trial. Ann Phys Rehabil Med. 2023 Jun;66(5):101765. doi: 10.1016/j.rehab.2023.101765. Epub 2023 Jun 2. PMID 37271020
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Schmidt M, Banzett RB, Raux M, Morelot-Panzini C, Dangers L, Similowski T, Demoule A. Unrecognized suffering in the ICU: addressing dyspnea in mechanically ventilated patients. Intensive Care Med. 2014 Jan;40(1):1-10. doi: 10.1007/s00134-013-3117-3. Epub 2013 Oct 17. PMID 24132382
- [Background] Rose L, Nonoyama M, Rezaie S, Fraser I. Psychological wellbeing, health related quality of life and memories of intensive care and a specialised weaning centre reported by survivors of prolonged mechanical ventilation. Intensive Crit Care Nurs. 2014 Jun;30(3):145-51. doi: 10.1016/j.iccn.2013.11.002. Epub 2013 Dec 3. PMID 24308899
- [Background] Hough CL, Steinberg KP, Taylor Thompson B, Rubenfeld GD, Hudson LD. Intensive care unit-acquired neuromyopathy and corticosteroids in survivors of persistent ARDS. Intensive Care Med. 2009 Jan;35(1):63-8. doi: 10.1007/s00134-008-1304-4. Epub 2008 Oct 23. PMID 18946661
- [Background] Kramer CL. Intensive Care Unit-Acquired Weakness. Neurol Clin. 2017 Nov;35(4):723-736. doi: 10.1016/j.ncl.2017.06.008. PMID 28962810